CLINICAL TRIAL: NCT04070885
Title: Cohort Follow-up: Progression and Consequences of Chronic Kidney Disease.
Acronym: NéphroTest
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2009/29
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Renal Diseases; Renal Function Disorder
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A dry tube of 7 ml of blood, two 4 ml ethylene-diamine-tetra-acetic acid tubes, a 4 ml heparinized tube and an 8.5 ml citrate dextrose acid tube will be collected from the patient.
  The urine will be taken from three 15 ml tubes.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sample — A dry tube of 7 ml of blood, two 4 ml EDTA tubes, a 4 ml heparinized tube and an 8.5 ml ACD-A tube will be collected from the patient.
Procedure: Urine sample — The urine will be taken from three 15 ml tubes.

SUMMARY:
This study aims to conduct a prospective collection of clinical and para-clinical data in patients with Chronic Renal Diseases to identify disease progression factors, markers of renal function, and the pathophysiology of Chronic Renal Diseases complications.

DETAILED DESCRIPTION:
Chronic Renal Diseases have a growing incidence and prevalence in France, with significant consequences in terms of morbidity and mortality, especially cardiovascular, and Public Health.

It is necessary to know better:

* the mechanisms leading to the progression of the Chronic Renal Diseases
* markers to quantify renal function and progression of the Chronic Renal Diseases
* the pathophysiology of Chronic Renal Diseases complications, cardiovascular, nutritional, or mineral metabolism in particular.

This study aims to conduct a prospective collection of clinical and para-clinical data in patients with Chronic Renal Diseases to identify disease progression factors, markers of renal function, and the pathophysiology of Chronic Renal Diseases complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Renal Disease, stage 2 to 5, non-dialysis patients over the age of 18,
* followed in the Nephrology Department of the Bordeaux University Hospital
* agreeing to participate in NephroTest
* affiliated with social security.

Exclusion Criteria:

* Patients under 18 years
* Patients with acute or rapidly progressive renal failure
* Patients with severe comorbidities or comorbidities that are life-threatening in the short term (<1 year)
* Patients who did not give their written consent to be included in the study
* Major incapacitated patients and psychiatric patients admitted to hospital

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participation in NephroTest will be offered to eligible patients by the doctors of the Nephrology Department, during consultations or as a result of hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2011-01-05 (Actual); Primary Completion 2015-03-20 (Actual); Study Completion 2015-03-20 (Actual)

PRIMARY OUTCOMES:
Estimated Glomerular Filtration Rate measurement | At 1 year after inclusion
  by isotope technique
Estimated Glomerular Filtration Rate measurement | At 2 year after inclusion
  by isotope technique
Measured Glomerular Filtration Rate | At 1 year after inclusion
  by isotope technique
Measured Glomerular Filtration Rate | At 2 years after inclusion
  by isotope technique

CONTACTS AND LOCATIONS:
Overall Officials: Christian COMBE, Pr, Principal Investigator — University Hospital, Bordeaux